CLINICAL TRIAL: NCT02854501
Title: Second Trimester Maternal Serum Homocysteine Levels and Uterine Artery Doppler for Prediction of Preeclampsia and Poor Placentation Disorders
Brief Title: Second Trimester Maternal Serum Homocysteine Levels and Uterine Artery Doppler for Prediction of Preeclampsia and Placentation Disorders
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Assistant professor, Cairo University
Other Study IDs: 153
Record Dates: First submitted 2016-08-01; First posted 2016-08-03 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Preeclampsia
Keywords: Homocysteine; Preeclampsia; poor placentation
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The plasma tHcy concentrations were measured by means of a fluorescence polarization immunoassay
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Uncomplicated pregnancies: women who did not develop any of the complications
- Preeclampsia: pregnant women who developed preeclampsia
- Isolated IUGR: participants were those who had IUGR
- Any complication: participants who developed other complications (abruptio placentae, stillbirth, or preterm labor).

SUMMARY:
The current study included the singleton pregnancies (without history of previous risk factors), had their homocysteine measured as part of a serum-screening program in addition to uterine artery Doppler. Sensitivity, specificity, positive and negative predictive values, for development of preeclampsia and other adverse pregnancy outcomes were assessed as follows; (1) Homocysteine cutoff level at 6.3 µmol/l; (2) Bilateral notches on Doppler with a mean RI >0.5, all unilateral notches with a mean RI >0.6, in addition, absence of notches with a mean RI >0.7; (3) Doppler assessment combined with the homocysteine cutoff (6.3 µmol/l).

DETAILED DESCRIPTION:
These participants had uterine artery Doppler investigations, as part of a routine scan between the 18th and the 22nd week of pregnancy. The investigators were blinded to the results of the biochemistry results.

All samples of the tHcy measurement were collected between 15 and 19 weeks of gestational age, as calculated from the last menstrual period or from early ultrasound dates (when the menstrual dates differed from the specified gestation). The plasma tHcy concentrations were measured by means of a fluorescence polarization immunoassay (9).

Uterine artery flow velocity waveforms were obtained using an SD 800 Doppler system (Philips Medical Systems, Gland, Switzerland) with a 3.5/5-MHz linear array probe. The high-pass filter was set at 100 Hz. One operator performed the measurements. The use of mean resistance index (RI) cutoff points with bilateral and unilateral notches has already been shown to improve the efficacy of uterine artery Doppler screening using qualitative assessment (10). A screen-positive or abnormal result was defined as bilateral notches and a mean RI >0.55 (50th centile), unilateral notches and a mean RI >0.65 (80th centile), and absence of notches and a mean RI >0.7 (95th centile) (11). Women with these abnormal results were offered growth scans, amniotic fluid volume assessment, and umbilical artery Doppler every 4 weeks until 36 weeks in view of the recognized increased risk of isolated IUGR (12), unless there were other clinical indications, which necessitated closer surveillance

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous pregnancies without history of previous risk factors for preeclampsia

Exclusion Criteria:

* multiple pregnancy, non-intact renal function, and hypertension before 20 weeks of gestation, diabetes mellitus and/or chronic diseases, women taking folic acid supplementations, women using antifolate drugs, and maternal age more than 40 years

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Spontaneous pregnancies without history of risk factors for preeclampsia were enrolled in the current study
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
development of placentation disorders | 28-40 weeks gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Kasr Alainy medical school

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Maged AM, Saad H, Meshaal H, Salah E, Abdelaziz S, Omran E, Deeb WS, Katta M. Maternal serum homocysteine and uterine artery Doppler as predictors of preeclampsia and poor placentation. Arch Gynecol Obstet. 2017 Sep;296(3):475-482. doi: 10.1007/s00404-017-4457-y. Epub 2017 Jul 8. PMID 28689278